CLINICAL TRIAL: NCT04313998
Title: Prevalence of Diabetes in Children and Its Risk Factors
Brief Title: The Effect of Early-life Risk Factors on the Etiology of Diabetes in Children: a Birth Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sijia Gu (Other)
Responsible Party: Sponsor-Investigator, Sijia Gu, Staff of Research Department, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: SCMCIRB-K2017021
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Umbilical cord blood and placenta were collected at birth,and parents' blood sample were collected on the first day after delivery

SUMMARY:
In recent years, with the rising prevalence of obesity among children, the incidence of type 2 diabetes in children and adolescents has continued to be increased. Some studies have found that impaired glucose metabolism appeared in 10-20% obese children. A large multicenter study project for children and adolescents showed that the prevalence of type 2 diabetes among children in the United States increased by 30.5% between 2001 and 2009. In addition, diabetes in children and adolescents, especially type 2 diabetes, has become more and more "younger". Diabetes appears in adolescence, which indicates that the damage of diabetes may come earlier, and it also has a significant impact on life quality and long-term survival. In recent years, more and more studies have shown that many adverse factors in the perinatal period would increase the risk of offspring suffering from metabolic diseases such as obesity and diabetes. Early life environmental factors would change the transcription and expression of obesity and diabetes-related genes through epigenetic regulation without changing the nucleotide sequence of the gene, then affecting the function of the gene and leading to diseases. Compared with the control group, pre-pregnant obese mothers and gestational diabetes mothers had higher DNA methylation levels in placenta leptin, which led to differences in the expression of leptin of offspring. A recent meta-analysis shows that the exposure to various social and environmental factors (diet, sleep, stress, bad habits, etc.) during pregnancy will affect the offspring. Due to the expression or methylation of CpG islands, these changes eventually lead to a variety of diseases including diabetes of offspring. However, most of previous researches mainly focused on the genetics or environmental factors. Meanwhile, most of the research focused on the Caucasian population. The differences between Asians and Westerners were few reported.

DETAILED DESCRIPTION:
Study Design: Prospective observational cohort study. Aim: To explore the effect of maternal sleep during pregnancy on offspring's growth and metabolism and the potential epigenetic mechanism.

Participants: Pregnant women with Gestational Diabetes Mellitus(GDM) and their children.

Study Procedure: Pregnant women with GDM were recruited during late pregnancy, and the children were followed up at birth, 42 days after birth, 3month, 6month, 12month, 18month and 24month. Demographic information, physical examination, developmental and psychiatric assessment, diet, and physical activity, as well as biological samples were collected for further study.

Collaborators on this study include: Renji hospital, affiliated shanghai jiaotong university school of medicine

ELIGIBILITY:
Inclusion Criteria:

* Long-term resident in Shanghai, and no relocation plan for 2 years
* Ultrasonography indicated singleton pregnancy at 34-36 weeks
* Willing to participate and be able to follow-up at the specified time
* Diagnosed with gestational diabetes mellitus

Exclusion Criteria:

* Preterm labor symptoms during pregnancy;
* Diagnosed gestational hypertension ;
* Diagnosed heart disease, liver and kidney disease.
* Apgar score was 7 or below at 1 minute or 5 minutes with history of asphyxia at birth or were admitted to the neonatal intensive care unit after birth.

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pregnant women with GDM were recruited during late pregnancy, and the children were followed up at birth, 42 days after birth, 3month, 6month, 12month, 18month and 24month.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Maternal sleep measured by Pittsburgh Sleep Quality Index(PSQI) | changes from late pregnancy,3 month, 6month, 9month, 12month, 18month, 24 month,36month,48month follow-up
  The PSQI total score represents the sum of component scores for subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medicine, and daytime dysfunction. A PSQI score >5 defined poor sleep quality. Higher scores implied lower sleep quality or more severe sleep disturbance.
Maternal sleep measured by Actiwatch | baseline
  Sleep assessment was a major part of the study. A 7-day assessment of mothers' sleep quality was conducted during the third trimester by using Actiwatch (AMI) and sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Children sleep measured by Actiwatch | changes from 3month,6month,12month ,18month and 24month follow-up
  Sleep assessment was a major part of the study. A 7-day assessment of mothers' sleep quality was conducted by using Actiwatch (AMI) and sleep diary. AMI is a sleep assessment system based on monitoring individual activity whose evaluation point is based on the sleep diary.
Childrens' anthropometrics | Changes from birth，42days, 3month,6month,12month ,18month and 24month follow-up
  Child weight and length/height as well as BMI (calculated by weight divided by the square of length/height) were obtained at each visit. Weight was measured using calibrated scales (Seca 335, Hamburg, Germany) and length was measured from the top of the head to the soles of feet using the same calibrated scale as weight. From 6 month，childrens' arm circumference, triceps and subscapular skinfold thicknesses were also measured.
Cord blood DNA methylation | at birth
  Cord blood samples were collected from the umbilical vein immediately after delivery, then were stored at 4 ℃ for a maximumof 4 h. They were then centrifuged, aliquoted, and stored in liquid nitrogen (-80℃) until assayed. DNA methylation was measured on bisulfite-converted genomic DNA in the company using the Illumina Infinium Human Methylation EPIC BeadChip (850k).
maternal metabolism index | baseline
  Leptin, Ghrelin, Adiponectin, Lipid profiles, Fasting glucose, Insulin-Like Growth Factor-1, Vitamin D, Ca, P, Fe, Ferritin, Transferrin were measured following a standard operating procedure.
infant metabolism index | baseline
  Leptin, Ghrelin, Adiponectin, Lipid profiles, Fasting glucose, Insulin-Like Growth Factor-1, Vitamin D, Ca, P, Fe, Ferritin, Transferrin were measured following a standard operating procedure.
paternal metabolism index | baseline
  Leptin, Ghrelin, Adiponectin, Lipid profiles, Fasting glucose, Insulin-Like Growth Factor-1, Vitamin D, Ca, P, Fe, Ferritin, Transferrin were measured following a standard operating procedure.
Children sleep measured by Brief Infant Sleep Questionnaire(BISQ) | changes from birth, 42days,3 month, 6month, 9month, 12month, 18month, 24 month follow-up
  Infant sleep problems reported by the mother and according to Brief Infant Sleep Questionnaire (BISQ). It is not a scale. The variables of the questionnaire included 1) nocturnal sleep duration (between the hours of 7 pm and 7 am); 2) daytime sleep duration (between the hours of 7 am and 7 pm); 3) number of night wakenings; 4) duration of wakefulness during the night hours (10 pm to 6 am); 5) nocturnal sleep-onset time (the time when the child falls asleep for the night); 6) settling time (latency to falling asleep for the night); 7) method of falling asleep; 8) location of sleep; 9) preferred body position; 10) age of child; 11) gender of child; 12) birth order; and 13) role of the responder who completed the BISQ. If the child woke up more than 3 times per night, spent more than 1 hour in wakefulness during the night, or spent less than 9 hours in sleep (day and night), then they were considered as poor sleepers.
Early Child Development | changes from 42days,3 month, 6month, 9month, 12month, 18month, 24 month follow-up
  The Griffiths Mental Development Scales (GMDS) assess the development of a child from 0 to 8 years across six separate subscales: Locomotor (A), Personal-social (B), Language (C), Eye-hand co-ordination (D), Performance (E), and Practical Reasoning (F).And the higher socres means better condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai children's medicial center affiliated shanghai jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China